CLINICAL TRIAL: NCT00898638
Title: Head and Neck Tumor Tissue Repository and Clinical Database
Brief Title: Tissue Sample Collection From Patients With Head and Neck Cancer and From Healthy Participants
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eben Rosenthal, Dept Chairperson Professor, Vanderbilt University Medical Center
Other Study IDs: CDR0000546682; P30CA068485 (NIH); VU-VICC-HN-0356; VU-VICC-IRB-030062
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I adenoid cystic carcinoma of the oral cavity; stage I basal cell carcinoma of the lip; stage I mucoepidermoid carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II basal cell carcinoma of the lip; stage II mucoepidermoid carcinoma of the oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III basal cell carcinoma of the lip; stage III mucoepidermoid carcinoma of the oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV basal cell carcinoma of the lip; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; recurrent basal cell carcinoma of the lip; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; recurrent squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9999 Days
Biospecimen Retention: Samples With DNA — Retrospective --Pathology archives will be reviewed and those with a sufficient amount of formalin-fixed tumor may be enrolled. Additionally, normal tissue from upper aerodigestive tract tissue excised for benign conditions will be collected. A one-time collection of medical data will be done for these cases. Specimens and datasets may also be incorporated from other studies with specimens and/or useful data left over.
  Prospective -- For non-tumor volunteers: After patient has signed consent, mouth cells and/or saliva samples will be obtained. If the patient agrees to having a biopsy, tissue may also be collected.
  For tumor patients: If the patient requires surgery, biological specimens will be collected day of surgery. The pathologist or designated lab personnel will oversee processing of the specimens. If the patient is scheduled to have a bronchoscopy, a bronchial washing may be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Non-tumor volunteers will be asked to participate at the time that they are attending a head and neck cancer screening clinic or at the time they are accompanying a patient to their appointment at the head and neck clinic. Intake sheets and biological specimens contributed by volunteers will be coded at the time of collection so that no identifiers are obtained. These specimens will not be linked to identifiers.
  Interventions: Other: biologic sample preservation procedure; Other: medical chart review
- Head and Neck Tumor patients: Eligible patients will be identified at the Vanderbilt Head & Neck Clinic by clinical and research staff. An appropriately trained staff member will discuss the protocol with the patient (including, risks, benefits, alternatives, etc.).
  Interventions: Other: biologic sample preservation procedure; Other: medical chart review

INTERVENTIONS:
Other: biologic sample preservation procedure
Other: medical chart review

SUMMARY:
RATIONALE: Collecting and storing samples of tissue, saliva, and blood from patients with cancer and from healthy participants to study in the laboratory may help the study of cancer in the future.

PURPOSE: This research study is collecting and storing tissue samples from patients with head and neck cancer and from healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Maintain and update a clinical database pertaining to diagnosis and treatment outcome of patients with head and neck cancer.
* Develop a repository of biospecimens from these patients.

OUTLINE: Tumor tissue samples and/or bronchial washings are collected from patients undergoing planned surgery and/or bronchoscopy, respectively. Buccal swabs and/or mouthwash samples and saliva samples are collected. Patients also undergo blood sample collection at baseline and then every 2-6 months thereafter.

Healthy participants contribute blood samples, buccal swabs, and mouthwash samples at baseline only.

Information about medical and family history and cancer risk factors is also collected.

PROJECTED ACCRUAL: No limit.

FOLLOW UP: Indefinite, until date of death or lost to follow up.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of head and neck cancer
  * Being treated at Vanderbilt University Medical Center for the cancer
  * Healthy participant

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Head and neck tumor patients, aged 18 and older and Healthy volunteers, aged 18 and older.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2003-02-13 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Maintenance of a clinical database pertaining to diagnosis and treatment outcome of patients with head and neck cancer | ongoing
  Collection of data for both groups from the Vanderbilt Otolaryngology Patient Intake questionnaire as well as the medical record, such as medical history, family history, and exposures to risk factors for cancer (tobacco and alcohol use), and results of tests related to diagnosis of tumor and treatment response (for tumor patients only).
Development of a repository of biospecimens | ongoing
  Collection of blood, tissue, saliva, bronchial washings and other specimens as indicated from both tumor and healthy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eben Rosenthal, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (4):
- United States (4):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No